CLINICAL TRIAL: NCT05129020
Title: Delivering Transcutaneous Auricular Neurostimulation as an Adjunct Treatment for Neonatal Opioid Withdrawal Syndrome
Brief Title: Neurostimulation to Improve NOWS Outcomes
Acronym: SPROUT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spark Biomedical, Inc. (Industry)
Collaborators: Medical University of South Carolina (Other); University of Texas Southwestern Medical Center (Other); University of Texas Health Science Center San Antonio (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBM-NOWS-02
Record Dates: First submitted 2021-11-04; First posted 2021-11-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Neonatal Opioid Withdrawal Syndrome; Neonatal Abstinence Syndrome
Keywords: auricular neurostimulation; vagus nerve stimulation; transcutaneous; withdrawal symptoms
MeSH Terms: conditions — Neonatal Abstinence Syndrome; Substance Withdrawal Syndrome

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized, double-blind, sham-controlled, multi-center, clinical trial in which neonates diagnosed with Neonatal Opioid Withdrawal Syndrome (NOWS) will be randomized 1:1 into one of two treatment groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each clinical site will have NICU nurses that will perform the Finnegan scale and be blind to the subjects' group designation. This will ensure a non-biased assessment of the Finnegan score, and importantly morphine dosing. Information regarding study intervention will be withheld from the blinded NICU nurses. NNNS assessors will also be blinded to information regarding study intervention to prevent biased NNNS scoring. All investigators will be blinded to subject treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active tAN + Morphine (Experimental)
  Interventions: Device: Sparrow Fledging Therapy System
- Sham tAN + Morphine (Sham Comparator)
  Interventions: Device: Sham Sparrow Fledging Therapy System

INTERVENTIONS:
Device: Sparrow Fledging Therapy System — tAN sessions will be administered up to four times per day for up to 20 days total. Active tAN will be set to run for 30 minutes one hour prior to each planned morphine dose. When the 30-minute tAN session is complete, the system will be turned off and unplugged.
  Arms: Active tAN + Morphine
Device: Sham Sparrow Fledging Therapy System — Participants randomized to the sham group will have the device earpiece applied at the same timepoints and for the same duration as the active group, but stimulation will not be turned on. tAN sessions will be administered up to four times per day for up to 20 days total. Sham tAN will be set to run for 30 minutes one hour prior to each planned morphine dose. When the 30-minute tAN session is complete, the system will be turned off and unplugged.
  Arms: Sham tAN + Morphine

SUMMARY:
The objective of this study is to determine if tAN therapy can reduce the median number of days of oral morphine administered to an infant after start of treatment.

DETAILED DESCRIPTION:
This study is designed as a randomized, double-blind, sham-controlled, multi-center, clinical trial in which neonates diagnosed with Neonatal Opioid Withdrawal Syndrome (NOWS) will be randomized 1:1 into one of two treatment groups:

1. Group 1: Active tAN + Morphine
2. Group 2: Sham tAN + Morphine

Morphine dosing for all infants will be managed by using the Finnegan Neonatal Abstinence Scoring System (FNASS), recorded every three hours.

After the participant exits the inpatient treatment phase of the study, they will enter the neurodevelopmental follow-up phase. The participant's parent or legal guardian will be contacted at 3, 9, 18, and 24 months of age to complete the Ages and Stages Questionnaire (ASQ-3) and the Sensory Profile 2 (SP-2). At 24 months, participants who fail in any sub-domain will be referred to their primary care physician for further neurodevelopmental assessment using the Bayley Scale of Infant and Toddler Development III (BSID-III) or other neurodevelopmental assessment.

ELIGIBILITY:
Inclusion Criteria

1. Neonates or infants >33 weeks gestational age with NOWS who have withdrawal scores requiring morphine replacement therapy
2. Clinically stable without respiratory support (exception for nasal cannula)
3. Congenital syndromes may be included if the infants do not have major, unrepaired anomalies

Exclusion Criteria

1. Unstable infants
2. Repeated episodes of autonomic instability (apnea or bradycardia) which are not self-resolving
3. Major unrepaired congenital anomalies impacting respiratory or cardiovascular system
4. Cardiomyopathy
5. Abnormal ear anatomy preventing the device to fit
6. Infants diagnosed with iatrogenic NOWS
7. Infants two weeks of age or older (after birth)
8. Neonates who have received more than 6 methadone doses or 24 hours of methadone dosing
9. Infants who are wards of the state
10. Participant has any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 33 Weeks to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Median number of days of oral morphine medication administered to the infant after start of active or sham tAN treatment. | Duration of morphine administration
Finnegan Neonatal Abstinence Scoring System (FNASS) | Day 1 - Day 30 (or day of discharge)
  Finnegan Neonatal Abstinence Scoring System (FNASS) is a validated assessment tool designed to measure 21 signs of withdrawal in infants. The tool provides a means to rate severity of withdrawal symptoms every three hours after feeding using a standard format.

SECONDARY OUTCOMES:
Median length of hospital stay due to NOWS | Through inpatient treatment phase completion, an average of one month
  Defined as the number of calendar days from first q3h opioid administration through the 48-hour observation period
Median length of hospital stay secondary to NOWS | Through inpatient treatment phase completion, an average of one month
  Defined as the number of calendar days from date of birth through date of discharge
Neonatal Neurobehavioral Scale (NNNS-II) | Baseline, Day 7, Day 15, and Day 30 (or day of discharge)
  The NNNS is a comprehensive and systematic assessment of an infant's response to a variety of items including handling, spontaneous behavior, motor activity and self-soothing as indicators of neurobehavioral performance. The NNNS examines neurobehavioral organization, neurological reflexes, motor development, active and passive tone, and signs of stress and withdrawal of the at-risk and drug-exposed infant. The NNNS document the range of withdrawal and stress behavior likely to be observed in intervention with substance-exposed infants. The scale consists of 13 domains: habituation, attention, arousal, regulation, handling procedures, quality of movement, excitability, lethargy, nonoptimal reflexes, asymmetric reflexes, hypertonicity, hypotonicity, and stress/abstinence scale. Summary scores are calculated and compared with percentile scores to determine how an infant compares with an at-risk sample. The NNNS has good psychometric properties and reliability.
Mean number of days of oral morphine medication administered | Day 1 - Day 30 (or day of discharge)
Mean number of days from birth to medical readiness for discharge | From day of birth through discharge, an average of one month
  Defined as the date where all of the following criteria are met: age of at least 96 hours, a period of at least 48 hours without receipt of an opioid, at least 24 hours without respiratory support and with 100% oral feeding, at least 24 hours from initiation of maximum caloric density

OTHER OUTCOMES:
Median length of time to reach oral morphine control dose | Day 1 - Day 30 (or day of discharge)
Mean total oral morphine delivered | Day 1 - Day 30 (or day of discharge)
Proportion of infants with episode(s) of bradycardia | Day 1 - Day 30 (or day of discharge)
Proportion of infants with episode(s) of apnea related to tAN | Day 1 - Day 30 (or day of discharge)
Proportion of infants with episode(s) of laryngospasms related to tAN | Day 1 - Day 30 (or day of discharge)
Neonatal Infant Pain Scale (NIPS) | Day 1 - Day 30 (or day of discharge)
  The Neonatal Infant Pain Scale (NIPS) is a validated pain scale utilized in the NICU. There are six components to the NIPS: facial expression, crying, breathing patterns, arm and leg movements, and state of arousal. The NIPS scale scoring ranges from 0-7, with scores greater than 3 indicating discomfort. A score of 3 is similar to the pain level associated with a heel stick procedure to obtain blood and the maximum score of 6 is similar to a circumcision procedure without analgesia. This measure will be taken immediately prior to, during, and after tAN therapy.
Number of infants with an Ages and Stages Questionnaire-3 (ASQ-3) Score greater than 2 standard deviations below the mean for any domain | At 3, 9, 18, and 24 months of age
  The ASQ-3 is a parent-completed developmental screening tool that pinpoints developmental progress in children between the ages of one month to 5 ½ years. The ASQ-3 is a series of 19 age-specific questionnaires screening communication, gross motor, fine motor, problem-solving, and personal adaptive skills; results in a pass/fail score for domains.
Number of infants who have scores outside of "typical performance", as calculated by a score greater than 1 standard deviation away from the mean, on the Sensory Profile 2 (SP-2) | At 3, 9, 18, and 24 months of age
  The SP-2 is a set of norm-referenced, parent and teacher questionnaires designed to assess the sensory processing patterns of children from birth through 14 years, 11 months. Information obtained from the Sensory Profile 2 helps identify ways sensory processing may be contributing to or interfering with a child's participation in home, school, and community. There are five different forms selected based on age: 1) Infant Sensory Profile 2 - Birth to 6 months; 2) Toddler Sensory Profile - 7 to 35 months; 3) Child Sensory Profile 2 - 3 to 15 years; 4) Short Sensory Profile 2 - 3 to 15 years; and 5) School Companion Sensory Profile 2 - 3 to 15 years. Each of the forms includes some combination of Sensory System, Behavioral, and Sensory Pattern scores.
Proportion of participants who do not meet criteria for normal neurodevelopment as measured by the Bayley Scale of Infant and Toddler Development III (BSID-III) or other neurodevelopmental assessment | At 24 months of age
  The BSID-III is an extensive formal developmental assessment tool for diagnosing developmental delays in early childhood. The BSID-III has three main subtests; the Cognitive Scale, the Language Scale, and the Motor Scale.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Medical University of South Carolina - Shawn Jenkins Children's Hospital, Charleston, South Carolina
  - UT Southwestern Medical Center / Parkland Memorial Hospital, Dallas, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
There is no plan to share participant data.

DOCUMENTS (1):
  • Informed Consent Form (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT05129020/ICF_001.pdf